CLINICAL TRIAL: NCT01570426
Title: Brain/Behavior Alterations in Pediatric Psychopathology
Brief Title: Brain Imaging and Computer Games in Children With Either Bipolar Disorder, ADHD, Anxiety or Healthy Controls
Acronym: BBPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bradley Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0195-07; K22MH074945 (NIH)
Record Dates: First submitted 2012-03-27; First posted 2012-04-04 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Bipolar Disorder; Attention Deficit Disorder With Hyperactivity; Attention Deficit Disorder Without Hyperactivity; Generalized Anxiety Disorder; Healthy
Keywords: Bipolar disorder; Mood disorders; ADHD; Attention Deficit Disorder with Hyperactivity; Attention Deficit Disorder without Hyperactivity; Anxiety disorders; Generalized anxiety disorder; Magnetic resonance imaging; Mental disorders; Mental disorders diagnosed in childhood; affective neuroscience; emotion; MRI; fMRI; neurocognitive tasks; imaging; Healthy controls; typical development
MeSH Terms: conditions — Bipolar Disorder; Attention Deficit Disorder with Hyperactivity; Generalized Anxiety Disorder; Mood Disorders; Anxiety Disorders; Mental Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Spit samples are collected for DNA/RNA extraction.Genetic tests will be performed at the Brown University affiliated Molecular Genetics Laboratory located at the Providence VA Medical Center. For privacy purposes, all genetic samples will be assigned a study code number to ensure that there is no identifiable information with them. After this study is over, genetic samples will be disposed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Bipolar Disorder: Children, 7- 17 years-old, who meet diagnostic criteria for bipolar disorder, Type 1
- ADHD/ADD: Children, 7-17 years-old, who meet diagnostic criteria for attention deficit/hyperactivity disorder (ADHD) OR attention deficit disorder (without hyperactivity)
- Generalized Anxiety Disorder (GAD): Children, 7-17 years-old, who meet diagnostic criteria for Generalized Anxiety Disorder (GAD)
- Health Controls: Children, ages 7-17 years-old, without a history of psychiatric diagnosis

SUMMARY:
The purpose of this research is to learn more about how children with mental health problems, including bipolar disorder (BD), attention deficit hyperactivity disorder (ADHD), and generalized anxiety disorder (GAD), differ from children without these problems. The investigators want to understand how these 4 groups of children differ in brain activity, function, and structure.

DETAILED DESCRIPTION:
This study has 2 visits (total time ~6 hours):

Visit #1 (2-3 hours), includes: (a) detailed description of study and study consent, (b) interviews about the child's mental health, mood, and behavior, and (c) a screening IQ test (word games, playing with blocks).

If a child fits our study criteria, they will play some special computer games, provide a spit sample for DNA, and parents/children will complete questionnaires.

All children fitting our study criteria, will also be invited to complete visit #2 (2 hours) consisting of a special MRI brain scan at Brown University (Providence, RI). To make sure all children feel comfortable in the MRI, they will spend time in our practice MRI (i.e., "MRI simulator") that looks and sounds just like the real MRI. During the actual MRI, children will play a computerized game in which they can win and lose points. The MRI lasts one and a half hours (at most).

Participants are compensated for their time.

ELIGIBILITY:
General Inclusion Criteria:

* English- speaking,children & adolescents between the ages of 7- 17
* consenting parent/guardian

General Exclusion Criteria:

* estimated IQ less than 70
* substance/alcohol use or dependence within the last 2 months
* Autism Spectrum Disorders or primary psychosis
* medical/neurological conditions that mimic the psychiatric disorders of interest
* implanted metal (NO BRACES or COCHLEAR IMPLANT)

For inclusion in the Bipolar group, participants:

* have to meet Diagnostic and Statistical Manual, 4th Edition Text Revision (DSM-IV-TR) criteria for BD Type I, including at least one lifetime episode of mania

For inclusion in the ADHD/ADD group, participants:

* meet DSM-IV-TR criteria for any subtype of ADHD or ADD
* can not currently meet diagnostic criteria for bipolar, depressive or anxiety disorders

For inclusion in the Generalized Anxiety Group (GAD), participants:

* have to meet DSM-IV-TR criteria for GAD
* can not currently meet diagnostic criteria for Obsessive Compulsive Disorder (OCD) or Post-Traumatic Stress Disorder (PTSD)

For inclusion in the Healthy Control group, participants:

* can not have a past/current history of psychiatric or substance use disorders
* can not have a first-degree relative (parents, brothers/sisters) with a history of psychiatric illness

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be recruited from in and around the Providence. Rhode Island area
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2007-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Behavioral performance on computerized tasks | Day 1
MRI data (neural activation) during behavioral task | Day 2
  structural, functional and diffusion tensor imaging data will be collected during the second day of the study.

SECONDARY OUTCOMES:
Genetic material | Day 1
  Genetic samples (spit sample) will be examined in relation to neural activation, function, and structure as well as behavioral performance on computerized tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States

REFERENCES:
- [Result] Dickstein DP, Gorrostieta C, Ombao H, Goldberg LD, Brazel AC, Gable CJ, Kelly C, Gee DG, Zuo XN, Castellanos FX, Milham MP. Fronto-temporal spontaneous resting state functional connectivity in pediatric bipolar disorder. Biol Psychiatry. 2010 Nov 1;68(9):839-46. doi: 10.1016/j.biopsych.2010.06.029. Epub 2010 Aug 24. PMID 20739018
- [Derived] Seymour KE, Pescosolido MF, Reidy BL, Galvan T, Kim KL, Young M, Dickstein DP. Emotional face identification in youths with primary bipolar disorder or primary attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2013 May;52(5):537-546.e3. doi: 10.1016/j.jaac.2013.03.011. PMID 23622855